CLINICAL TRIAL: NCT05094206
Title: Phase I Trial of Anti-CD20, Anti-CD19, Anti-CD22 CAR (CAR20.19.22) T-cells for Relapsed, Refractory B-cell Malignancies
Brief Title: CAR20.19.22 T-cells in Relapsed, Refractory B-cell Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Treated four patients: 2 at a dose of 1x10^6 cells/kg and 2 ad at dose of 2.5x10^6 cells/kg. All four patients had no in-vivo expansion and no meaningful response to therapy. At this point per FDA guidance we will not be treating more patients.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Miltenyi Biotec, Inc. (Industry)
Responsible Party: Principal Investigator, Nirav Shah, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00041528
Record Dates: First submitted 2021-10-17; First posted 2021-10-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: B-cell Non Hodgkin Lymphoma; B-cell Chronic Lymphocytic Leukemia
Keywords: B-cell antigens; B-cell Non Hodgkin Lymphoma; B-cell Chronic Lymphocytic Leukemia; CAR-T; Chimeric antigen receptor T-cell therapy; CAR Therapy
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Indolent B-cell NHL Dose Level -2: 0.75x10^6 cells/kg: CAR20.19.22 (Experimental): The investigators will start at a dose of 2.5x10^6 cells/kg and either escalate or de-escalate based on the presence of toxicities.
  Interventions: Biological: 0.75x10^6 cells/kg CAR20.19.22 cells
- Indolent B-cell NHL Dose Level -1: 1x10^6 cells/kg: CAR20.19.22 (Experimental): The investigators will start at a dose of 2.5x10^6 cells/kg and either escalate or de-escalate based on the presence of toxicities.
  Interventions: Biological: 1x10^6 cells/kg CAR20.19.22 cells
- Indolent B-cell NHL Dose Level 0: 2.5x10^6 cells/kg: CAR20.19.22 (Experimental): The investigators will start at a dose of 2.5x10^6 cells/kg and either escalate or de-escalate based on the presence of toxicities.
  Interventions: Biological: 2.5x10^6 cells/kg CAR20.19.22 cells
- Indolent B-cell NHL Dose Level 1: 5x10^6 cells/kg: CAR20.19.22 (Experimental): The investigators will start at a dose of 2.5x10^6 cells/kg and either escalate or de-escalate based on the presence of toxicities.
  Interventions: Biological: 5x10^6 cells/kg CAR20.19.22 cells
- Indolent B-cell NHL Dose Expansion: CAR20.19.22 (Experimental): The maximum tolerated dose intervention will be updated when it is determined. It will be one of four doses: 0.75x10^6 cells/kg, 1x10^6 cells/kg, 2.5x10^6 cells/kg or 5x10^6 cells/kg.
  Interventions: Biological: Dose expansion: The maximum tolerated dose of CAR20.19.22 cells
- Aggressive B-cell NHL Dose Level -1: .75x10^6 cells/kg: CAR20.19.22 (Experimental): The investigators will start at a dose of 1x10^6 cells/kg and either escalate or de-escalate based on the presence of toxicities.
  Interventions: Biological: 0.75x10^6 cells/kg CAR20.19.22 cells
- Aggressive B-cell NHL Dose Level 0: 1x10^6 cells/kg: CAR20.19.22 (Experimental): The investigators will start at a dose of 1x10^6 cells/kg and either escalate or de-escalate based on the presence of toxicities.
  Interventions: Biological: 1x10^6 cells/kg CAR20.19.22 cells
- Aggressive B-cell NHL Dose Level 1: 2.5x10^6 cells/kg: CAR20.19.22 (Experimental): The investigators will start at a dose of 1x10^6 cells/kg and either escalate or de-escalate based on the presence of toxicities.
  Interventions: Biological: 2.5x10^6 cells/kg CAR20.19.22 cells
- Aggressive B-cell NHL Dose Level 2: 5x10^6 cells/kg: CAR20.19.22 (Experimental): The investigators will start at a dose of 1.0x10^6 cells/kg and either escalate or de-escalate based on the presence of toxicities.
  Interventions: Biological: 5x10^6 cells/kg CAR20.19.22 cells
- Aggressive B-cell NHL Dose Expansion: CAR20.19.22 (Experimental): The maximum tolerated dose intervention will be updated when it is determined. It will be one of four doses: 0.75x10^6 cells/kg, 1x10^6 cells/kg, 2.5x10^6 cells/kg or 5x10^6 cells/kg.
  Interventions: Biological: Dose expansion: The maximum tolerated dose of CAR20.19.22 cells

INTERVENTIONS:
Biological: 0.75x10^6 cells/kg CAR20.19.22 cells — Dose escalation: CAR20.19.22 cells will be administered at one of three dose levels either fresh or thawed after cryopreservation by IV injection.
  Dose expansion: The maximum tolerated dose intervention will be updated when it is determined. It will be one of four doses: 0.75x10^6 cells/kg, 1x10^6 cells/kg, 2.5x10^6 cells/kg or 5x10^6.
  Arms: Aggressive B-cell NHL Dose Level -1: .75x10^6 cells/kg: CAR20.19.22; Indolent B-cell NHL Dose Level -2: 0.75x10^6 cells/kg: CAR20.19.22
Biological: 1x10^6 cells/kg CAR20.19.22 cells — CAR20.19.22 cells will be administered at one of four dose levels either fresh or thawed after cryopreservation by IV injection.
  Dose expansion: The maximum tolerated dose intervention will be updated when it is determined. It will be one of four doses: 0.75x10^6 cells/kg, 1x10^6 cells/kg, 2.5x10^6 cells/kg or 5x10^6.
  Arms: Aggressive B-cell NHL Dose Level 0: 1x10^6 cells/kg: CAR20.19.22; Indolent B-cell NHL Dose Level -1: 1x10^6 cells/kg: CAR20.19.22
Biological: 2.5x10^6 cells/kg CAR20.19.22 cells — CAR20.19.22 cells will be administered at one of four dose levels either fresh or thawed after cryopreservation by IV injection.
  The maximum tolerated dose intervention will be updated when it is determined. It will be one of four doses: 0.75x10^6 cells/kg, 1x10^6 cells/kg, 2.5x10^6 cells/kg or 5x10^6.
  Arms: Aggressive B-cell NHL Dose Level 1: 2.5x10^6 cells/kg: CAR20.19.22; Indolent B-cell NHL Dose Level 0: 2.5x10^6 cells/kg: CAR20.19.22
Biological: 5x10^6 cells/kg CAR20.19.22 cells — CAR20.19.22 cells will be administered at one of four dose levels either fresh or thawed after cryopreservation by IV injection.
  The maximum tolerated dose intervention will be updated when it is determined. It will be one of four doses: 0.75x10^6 cells/kg, 1x10^6 cells/kg, 2.5x10^6 cells/kg or 5x10^6.
  Arms: Aggressive B-cell NHL Dose Level 2: 5x10^6 cells/kg: CAR20.19.22; Indolent B-cell NHL Dose Level 1: 5x10^6 cells/kg: CAR20.19.22
Biological: Dose expansion: The maximum tolerated dose of CAR20.19.22 cells — Dose expansion: The maximum tolerated dose intervention will be updated when it is determined. It will be one of four doses: 0.75x10^6 cells/kg, 1x10^6 cells/kg, 2.5x10^6 cells/kg or 5x10^6 cells/kg.
  Arms: Aggressive B-cell NHL Dose Expansion: CAR20.19.22; Indolent B-cell NHL Dose Expansion: CAR20.19.22

SUMMARY:
In this phase I study, the investigators will first evaluate the safety of CAR20.19.22 T-cells in patients with B-cell non-Hodgkin lymphoma (NHL) / chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
This is a phase I, interventional, open label, dose-finding treatment study designed to evaluate the safety and efficacy CAR20.19.22 T-cells in adult patients with B-cell malignancies that have failed prior therapies.

ELIGIBILITY:
Inclusion Criteria for B-cell for non-Hodgkin lymphoma (NHL) and CLL (chronic lymphocytic leukemia) patients

1. Patients must be aged ≥18 years to 80 years with relapsed or refractory B-cell non-Hodgkin Lymphoma or chronic lymphocytic leukemia.
2. Absolute CD3 count ≥50 mm^3.
3. MRI brain and lumbar puncture with cerebrospinal fluid (CSF) analysis by cytology and flow cytometry without evidence of central nervous system (CNS) involvement ONLY in patients with history of CNS involvement or clinical suspicion at the time of enrollment.
4. Measurable disease must be documented within 4 weeks of apheresis date and is defined as nodal lesions >15 mm in the long axis or extranodal lesions >10 mm in long OR bone marrow involvement that is biopsy proven.
5. Karnofsky performance score ≥70.
6. Adequate hepatic function, defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase < 3x upper limit of normal (ULN); serum bilirubin < 2.0 mg/dL
7. ANC≥1000 with no G-CSF within 72 hours or pegylated G-CSF within 10 days unless bone marrow involvement is present.
8. Platelets ≥ 50,000 with no transfusion within 72 hours of eligibility testing unless bone marrow involvement is present.
9. Adequate renal function, defined as creatinine clearance≥60 ml/min AND serum Cr≤1.5 mg/dL.
10. Able to provide written informed consent.
11. Agree to practice birth control during the study.
12. Adequate cardiac function as indicated by New York Heart Association (NYHA) classification I or II AND left ventricular ejection fraction of ≥45% (by cardiac echocardiogram (ECHO) or MUGA) and adequate pulmonary function as indicated by room air oxygen saturation of ≥90%.
13. Expected survival >12 weeks.
14. Negative urine or serum pregnancy test in females of childbearing potential at study entry.
15. Meet criteria for regarding fertility and contraception detailed below.
16. No contraindication to central line access.
17. Diagnosis of CLL or B-cell NHL including follicular lymphoma, marginal zone lymphoma (splenic, nodal, extranodal), mantle cell lymphoma, Burkitt lymphoma, and DLBCL with associated subtypes (high-grade or aggressive B-cell lymphoma, T-cell/histocyte rich B-cell lymphoma, primary mediastinal B-cell lymphoma, Epstein-Barr virus (EBV) + diffuse large B-cell lymphoma, transformed lymphoma such as transformed follicular or marginal zone, and Richter's transformation).
18. For CLL patients, must have active, measurable disease (>5% CLL involvement of marrow or nodal disease as noted above) and failed/progressed or been intolerant to both covalent Bruton's tyrosine kinase (BTK) inhibitors (ibrutinib, acalabruinitib, or zanabrutinib) and B-cell lymphoma 2 (BCL2) inhibitors (e.g., venetoclax).
19. For B-cell NHL patients must have active, measurable disease as defined in Inclusion criteria #4, relapsed or refractory disease within 12 months of their last lymphoma directed treatment. Additionally patient must meet, and meet the following criteria as applicable:

    1. Patients who relapsed within 12 months of autologous stem cell transplant or allogeneic stem cell transplant and have measurable disease are eligible.
    2. For patients who have not had a prior autologous/allogeneic transplant they must have received an anti-CD20 monoclonal antibody and at minimum two prior treatment regimens. ONE of the regimens must include a disease appropriate regimen as listed below:

    i. For large cell or Burkitt lymphoma: anthracycline containing treatment (e.g., rituximab, cyclophosphamide, doxorubicin hydrochloride (hydroxydaunorubicin), vincristine sulfate (Oncovin), and prednisone (R-CHOP), R-EPOCH, HyperCVAD, Pola-R-CHP, etc.).

ii. For follicular lymphoma: either prior bendamustine or anthracycline based therapy.

iii. For mantle cell lymphoma: either prior bendamustine, anthracycline based regimen, or cytarabine based therapy.

iv. For marginal zone lymphoma: prior bendamustine based therapy.

Exclusion Criteria for ALL patients.

1. Positive beta-human chorionic gonadotropin (HCG) in female of child-bearing potential.
2. Confirmed active human immunodeficiency virus (HIV), Hepatitis B or C infection.
3. History of significant autoimmune disease OR active, uncontrolled autoimmune phenomenon requiring steroid therapy defined as >20 mg of prednisone or equivalent daily.
4. Presence of ≥grade 3 non-hematologic toxicities as per CTCAE version 5.0 from any previous treatment unless it is felt to be due to underlying disease.
5. Concurrent use of investigational therapeutic agents or enrollment on another therapeutic clinical trial at any institution. Minimum of 14 days or 5 half-lives of the drug (whichever is shorter) washout prior to apheresis.
6. Refusal to participate in the long-term follow-up protocol.
7. Patients with active CNS involvement by malignancy on MRI or by lumbar puncture.

   a. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was >4 weeks before enrollment and a remission documented within 8 weeks of planned CAR T-cell infusion by MRI brain and CSF analysis.
8. Previous recipients of allogeneic hematopoietic stem cell transplantation (AHCT) are excluded if they are <100 days' post-transplant, have evidence of active graft-versus-host-disease (GVHD) of any grade, or are currently on immunosuppression.
9. Anti-CD20 directed treatment within 4 weeks of cell infusion.
10. Anti-CD19 directed treatment within 4 weeks of cell infusion.
11. Anti-CD22 directed treatment within 4 weeks of cell infusion.
12. Cytotoxic chemotherapy, oral chemotherapeutic agents or antibody directed treatment within 14 days of lymphodepletion.

    1. Radiation is allowed to a single symptomatic site as long as other sites of measurable disease are present on eligibility scan.
    2. If patients receive steroids or any systemic disease targeting treatment, repeat scans are needed to confirm disease burden pre-lymphodepletion.
13. Cytotoxic chemotherapy, oral chemotherapeutic agents or antibody directed treatment within 14 days of apheresis.

    a. Corticosteroids are allowable up until 7 days prior to apheresis.
14. Patients post solid organ transplant who develop high grade lymphomas or leukemias.
15. Concurrent active malignancy other than basal or squamous cell carcinomas of the skin.
16. Prior CAR T-cell therapy (autologous or allogeneic) unless >90 days from prior CAR with repeat biopsy post-CAR demonstrating CD19 or CD20 expression of ≥20%.

Special Criteria for regarding Fertility and Contraception:

Female subjects of reproductive potential (women who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone a sterilization procedure [hysterectomy or bilateral oophorectomy]) must have a negative serum or urine pregnancy test performed as part of eligibility criteria. Lactating women are eligible for this study but will be asked to not provide breast milk to their child from Day -4 through Day +90 after CAR T-cell therapy. It is possible they may no longer be able to lactate after receiving chemotherapy and treatment.

Due to the high-risk level of this study, while enrolled, all subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). Additionally, if participating in sexual activity that could lead to pregnancy, the study subject must agree to use reliable and double barrier methods of contraception during the follow-up period of the protocol.

Acceptable birth control includes a combination of two of the following methods:

* Condoms (male or female) with or without a spermicidal agent.
* Diaphragm or cervical cap with spermicide.
* Intrauterine device (IUD).
* Hormonal-based contraception.

Subjects who are not of reproductive potential (women who are premenarche or have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy tubal ligation, salpingectomy, and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Number of Non-hematologic Adverse Events after Infusion | 28 days after infusion
  Occurrence of adverse events will be defined as non-hematologic Grade 3/4 toxicity grade per NCI CTCAE version 5.0.
Number of grade 3-4 cytokine release syndrome (CRS). | 28 days after infusion
  Grade 3-4 CRS as graded per the recent Transplant and Cell Therapy (TCT) consensus criteria.
Number of grade 3-4 immune effector cell-associated neurotoxicity syndrome (ICANS) | 28 days after infusion
  Grade 3-4 ICANS as graded per the recent Transplant and Cell Therapy (TCT) consensus criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Shah, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin and Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No